CLINICAL TRIAL: NCT07158723
Title: Assessing the Role of Higher Protein Diets in Managing Metabolic Complications of Polycystic Ovary Syndrome (PCOS)
Brief Title: Protein and Polycystic Ovary Syndrome (PCOS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas, Fayetteville (Other)
Collaborators: Arkansas Biosciences Institute (Unknown)
Responsible Party: Principal Investigator, Jamie Baum, Associate Professor, University of Arkansas, Fayetteville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2503592283
Record Dates: First submitted 2025-08-19; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Polycystic Ovary Syndrome (PCOS)
Keywords: PCOS; polycystic ovary syndrome; protein; women; wellbeing; metabolism
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Caloric Restriction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Calorie restricted control (Active Comparator)
  Interventions: Other: Calorie restriction
- Control and Protein (Active Comparator)
  Interventions: Other: Higher protein dietary pattern
- Calorie restricted PCOS (Active Comparator)
  Interventions: Other: Calorie restriction
- PCOS Protein (Active Comparator)
  Interventions: Other: Higher protein dietary pattern

INTERVENTIONS:
Other: Higher protein dietary pattern — Follow energy-restricted (10% calorie reduction), higher protein dietary pattern (1.6 g protein/kg body weight)
  Arms: Control and Protein; PCOS Protein
Other: Calorie restriction — Follow energy-restricted (10% calorie reduction) dietary pattern for 16 weeks. No restrictions on macronutrient content.
  Arms: Calorie restricted PCOS; Calorie restricted control

SUMMARY:
Polycystic ovary syndrome (PCOS) is a significant public health problem and is one of the most common hormonal disturbances affecting women of reproductive age. Women with PCOS are often insulin resistant, increasing their risk for cardiometabolic health problems (e.g., type 2 diabetes, heart disease, high blood pressure, sleep apnea, anxiety, depression, and stroke) especially if they are overweight. Lifestyle modifications, including dietary changes and regular physical activity, may alleviate metabolic dysfunction in women with PCOS and are often the first line of management for patients with PCOS. Several studies have identified protein as a key nutrient for regulation of energy balance, maintenance of skeletal muscle mass, and improving cardiometabolic health across the lifespan. However, the effect of increased protein intake (30% of total energy intake) on cardiometabolic health in women with PCOS has not been well-defined and mechanisms for these effects have not been identified.

There is an evident need for well-designed, randomized controlled trials evaluating the efficacy of increased protein intake in women with PCOS on markers of cardiometabolic health. Preliminary data from collaborative projects with the investigators on this proposal suggest that increasing protein in the diet has the potential to improve markers of cardiometabolic health, potentially through improvements in body composition and/or changes in cortisol, energy metabolism, inflammation, and neurological regulators

ELIGIBILITY:
Inclusion Criteria:

* Females ages 18-50 years
* Confirmed diagnosis of PCOS
* Body mass index (BMI) between 18.5 and 35 kg/m2
* Stable body weight for at least 3 months (+ 5 pounds)
* Willingness to consume both plant- and animal-based protein meals

Exclusion Criteria:

* Smoking or use of nicotine products
* Smoking, vaping, and/or use of marijuana products
* More than 4 alcoholic beverages per week
* Food allergies or dietary restrictions incompatible with test meals
* Diagnosed diabetes (type 1 or 2) or other preexisting chronic disease(s).
* Use of medications that interfere with study outcomes (e.g., metformin, GLP-1 agonists, etc.)
* Consumption of more than 0.8 g/protein/kg body weight
* Underweight
* Taking nutritional supplements

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-03 (Estimated)

PRIMARY OUTCOMES:
Lean body mass | 0 and 16 weeks.
  Lean body mass will be measured using dual x-ray absorptiometry.

SECONDARY OUTCOMES:
Body fat mass | 0 and 16 weeks
  Total body fat and body fat distribution will measured using dual x-ray absorptiometry.
Sleep Duration | Sleep will be measured every 8 weeks (0, 8, and 16 weeks)
  Sleep quality and duration will be assessed objectively via an ActiGraph triaxial wrist accelerometer GT3X+, ActiGraph, LLC, Pensacola, FL, USA), a validated method of sleep assessment. Each participant will wear an ActiGraph monitor on the non-dominant wrist for 24-hour per day for seven days (except when bathing or involved in water activities) prior to the start of the intervention, 8-, and 16-weeks. Actigraphs will be fitted securely on each participants wrist. Participants will receive sleep diaries to define "time in bed" and "time out of bed". Researchers will use the indicated "start" and "end" points to define a sleep region to be analyzed within the ActiGraph software. Sleep outcomes will be calculated based on epoch-to-epoch sleep/wake algorithms within the defined sleep period. Data were processed by using the ActiLife Version 6.9.2 software (Pensacola, FL, USA) and sleep will be scored via the Cole-Kripke algorithm.
Mood | Every 4 weeks (0, 4, 8, 12, 16 weeks)
  The Profile of Mood States (POMS) questionnaire consists of 65 questions containing a one-word adjective of mood to measure and identify six affective states. The six identifiable mood/affective states are tension-anxiety, depression-dejection, anger-hostility, vigor-activity, fatigue/-inertia, and confusion-bewilderment. Participants will be instructed to define their mood on a 5-point Likert scale ranging from 0 to 4. The numbers refer to the following descriptive phrases: 0 = Not at all, 1 = A little, 2 = Moderately, 3 = Quite a bit, 4 = Extremely. To obtain the score for reach identifiable mood/affective state subscale, the sum of the responses for each adjective is calculated. The subscale scores range from 0 up to 36, 60, 48, 32, 28, and 28 for tension-anxiety depression-dejection, anger-hostility, vigor-activity, fatigue/-inertia, and confusion-bewilderment respectively. Higher subscale scores for all affect states, but the vigor domain represent poorer mood.
Quality of Life perception | Every 4 weeks (0, 4, 8, 12, and 16 weeks)
  Health-related quality of life will be assessed using the 36-Item Short Form Health Survey (SF-36). The instrument consists of 36 items grouped into eight domains: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health. Items will be scored using standard Likert-type response scales and coded according to established procedures. Raw scores for each domain were summed and linearly transformed to a 0-100 scale, with higher scores indicating better health status.
Energy expenditure | Every 4 weeks (0, 4, 8, 12 and 16 weeks)
  Indirect calorimetry will be used to measure energy expenditure
Plasma amino acid concentrations | Every 4 weeks (0, 4, 8, 12 and 16 weeks).
  Plasma amino acids will be measured using UPL.
Inflammatory biomarkers | Every 4 weeks (0, 4, 8, 12, and 16 weeks).
  Inflammatory status will be evaluated using established circulating biomarkers that reflect systemic, low-grade inflammation. The primary analytes include high-sensitivity C-reactive protein (hs-CRP), interleukin-6 (IL-6), and tumor necrosis factor-alpha (TNF-α). hs-CRP is an acute-phase reactant produced by the liver and is widely used as a sensitive indicator of chronic inflammation and cardiovascular risk. IL-6 is a pro-inflammatory cytokine that plays a central role in immune regulation and metabolic function, while TNF-α is a key mediator of systemic inflammation and tissue catabolism. Together, these biomarkers provide complementary information on both acute-phase and cytokine-mediated pathways of inflammation and are commonly used in clinical and epidemiological studies to quantify inflammatory burden.
Subjective Sleep Measurements | Subjective sleep will be measured at 0, 4, 8, 12, and 16 weeks.
  Subjective measure of sleep quality will be assessed via the Pittsburgh Sleep Quality Index (PSQI) . The 19-item PSQI questionnaire addresses seven components of subjective sleep quality: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medications, and daytime dysfunction. In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global sleeping score (GSS) with a range of 0 to 21. Higher scores indicate worse sleep quality. A compiled global score of the seven scored components distinguishes good sleepers (≤ 5) from poor sleepers (>5). According to a test-retest reliability and validity experiment, as a marker for sleep disturbances, a PSQI GSS > 5 has a sensitivity of 98.7 and specificity of 84.4.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Human Nutrition, Fayetteville, Arkansas, United States

IPD SHARING:
Plan to Share IPD: Undecided